CLINICAL TRIAL: NCT03942744
Title: Molecular Mechanisms Involved in Cell Adhesion and Migration Process: Effect of Treatment of Chronic Kidney Disease on Endothelial Dysfunction
Brief Title: The Effect of High-flux Hemodialysis and On-line Hemodiafiltration on Endothelial Function.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Alejandro Martin-Malo, Professor of Medicine Chief of Dialysis Unit, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PI17/01785
Record Dates: First submitted 2019-03-05; First posted 2019-05-08 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Hemodialysis; Endothelial dysfunction; Atherogenesis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Intervention Model Description: prospective randomized crossover study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-flux hemodialysis (No Intervention): high-flux hemodialysis cut-off membrane above 50
- on-line hemodiafiltration (Active Comparator): postdilutional on-line hemodiafiltration with a convective transport above 21 liters
  Interventions: Device: on-line hemodiafiltration

INTERVENTIONS:
Device: on-line hemodiafiltration — on-line postdilutional hemodiafiltration with high convective transport above 21 liters
  Arms: on-line hemodiafiltration

SUMMARY:
The main aim of this project is to evaluate, in patients with chronic kidney disease (CKD5D), the role of adhesion molecules in leukocyte adhesion and transendothelial migration involved in atherogenesis. This trial is a prospective randomized crossover study in CKD5D hemodialysis patients followed in the Nephrology Unit of the Reina Sofia University Hospital (Cordoba, Spain). The estimated inclusion period is two years, with a follow-up of 24 months. Patients will be randomized to high-flux hemodialysis versus online hemodiafiltration with high convective transport (above 21 liters); after 6 months in each dialysis modality they will be switched the other technique for another 6 months. Then, patients will be maintained during 4 weeks in conventional hemodialysis "wash out period", before being started in the other dialysis modality.

DETAILED DESCRIPTION:
The main aim of this project is to evaluate, in patients with chronic kidney disease (CKD5D), the role of adhesion molecules in leukocyte adhesion and transendothelial migration involved in atherogenesis. This trial is a prospective randomized crossover study in CKD5D hemodialysis patients followed in the Nephrology Unit of the Reina Sofia University Hospital (Cordoba, Spain). The estimated inclusion period is two years, with a follow-up of 24 months. Patients will be randomized to high-flux hemodialysis versus online hemodiafiltration with high convective transport (above 21 liters); after 6 months in each dialysis modality they will be switched the other technique for another 6 months. Then, patients will be maintained during 4 weeks in conventional hemodialysis "wash out period", before being started in the other dialysis modality. Patients will be stratified by age, gender and the presence of diabetes. Routine analytical determinations (urea, creatinine, sodium, potassium, chlorine, total CO2, calcium, phosphorus, FA, PTH, levels 25OH, β2m, ALT, hemoglobin, leukocytes, platelets, glucose, uric acid, total proteins, albumin , PCR, IL-6, ferritin, TSAT and homocysteine), characteristics of hemodialysis and dialysis dose (Kt / V and Kt) will be recorded. Residual renal function will be analysed every three months. In plasma, microRNAs profile and FGF23 levels will be determined. Markers of endothelial dysfunction (CD31 +, CD41-, CD144, CD62E) and subclinical atherosclerosis markers (CD11b, CD41 +) will be measured. The hospitalization and mortality rate due to cardiovascular causes and concurrent cardiovascular events throughout the study (acute myocardial infarction, stroke, transient ischemic attack and peripheral vascular disease) will be assessed along the study period.

ELIGIBILITY:
Inclusion Criteria:

* Vascular access with a blood flow > 300ml/min
* Age >18 <80 years written informed consent

Exclusion Criteria:

* Neoplasia
* B hepatitis
* Acute or chronic inflammation life expectance less than one year Included in living donor transplant list immunosupressive drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Effect of two different dialysis modalities (high flux vs online hemodiafiltration) on endothelial function markers: CD31,CD41,CD34; as measured by the percent of labeled cells obtained by flow cytometry. | 6 months
  These parameters will assessed, in patients with chronic kidney disease (CKD5D), Blood will be drawn before the dialysis session following the scheduled of the protocol. The measuremets of CD31 CD41 CD34 will be performend by flow cytometry according to the standard methodology described in methods.

SECONDARY OUTCOMES:
Effect of two different dialysis modalities ( high flux vs online hemodiafiltration) on hospitalization (hospital admission days/year). | 6 months
  Effect of two different dialysis modalities ( high flux vs online hemodiafiltration) on hospitalization (hospital admission days/year). Cardiovascular causes and concurrent cardiovascular events throughout the study (acute myocardial infarction, stroke, transient ischemic attack and peripheral vascular disease) will be also recorded throughout the study.
Effect of two different dialysis modalities ( high flux vs online hemodiafiltration) on Serum concentration of Fibroblast Growth Factor FGF23 (pg/ml) . | 6 months
  The serum concentration of Fibroblast Growth Factor FGF23 will be quantified using commercially available ELISA Kit. (pg/ml). Blood samples will be obtained before the dialysis session.
Effect of two different dialysis modalities ( high flux vs online hemodiafiltration) on vascular injury related microRNAs (relative expression) | 6 months
  The relative expression of microRNAs (126-3p, 223-3p,363-3p, 191-5p). will be determined by RTq-PCR. Blood samples will be obtained before the dialysis session.

CONTACTS AND LOCATIONS:
Overall Officials: alejandro martin-malo, MD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba
Locations (2):
- Spain (2):
  - Hospital universitario Reina Sofia, Córdoba, Cordoba
  - Alejandro Martinmalo, Córdoba, Córdoba

IPD SHARING:
Plan to Share IPD: Yes
The individual data will be available in this report after deidenttification (text, tables, figures and appendices) to those researchers who provide a methodologically sound proposal and for meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after the end of the study until one year the article publication.
Access Criteria: To obtain the data, a proposal must be sent to uicec@imibic.org. To gain access, data requestors will need to sign a data access agreement.